CLINICAL TRIAL: NCT03541473
Title: Assessment of Nutrition on Brain Energy Metabolism in Humans Aged 50+: Measurement of Phosphate Metabolites by 31P-MRS
Brief Title: Phosphate Metabolites in Brain of Humans Aged 50+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: Ecole Polytechnique Fédérale de Lausanne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17.20.BIO
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Basic Science

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peptamen® 1.5 Vanilla (Active Comparator)
  Interventions: Dietary Supplement: Peptamen® 1.5 Vanilla
- Boost Plus® Vanilla (Placebo Comparator)
  Interventions: Dietary Supplement: Boost Plus® Vanilla

INTERVENTIONS:
Dietary Supplement: Peptamen® 1.5 Vanilla — Nutritionally complete formula with 10g MCT in 250 mL, commercially available
  Arms: Peptamen® 1.5 Vanilla
Dietary Supplement: Boost Plus® Vanilla — Product of same nutritional composition but without MCT
  Arms: Boost Plus® Vanilla

SUMMARY:
The objective of this research project is to determine in elderly subjects (>50 year old) by 31P-MRS the brain concentration of phosphorous metabolites species and fluxes, before and after consumption of 2 commercially available oral nutrition products

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 50 and 75 years
* Healthy, based on the medical screening visit
* Normal BMI for age (18.5-29.9 kg/m2)
* Able to understand and to sign a written informed consent prior to trial entry
* Informed consent signed

Exclusion Criteria:

* Known type 1 or type 2 diabetes, on anamnesis
* Family history of type 2 diabetes (parents)
* Any other metabolic disease possibly impacting the postprandial glucose and insulin response (on anamnesis, to the opinion of the medical expert)
* Malabsorptive disorders including but not limited to pancreatitis, Crohn's disease, etc, to the opinion of the medical expert
* Any ongoing medication impacting dietary fat absorption and metabolism like statins, bile acid sequestrants, lipid lowering medications, or fibrates , to the opinion of the medical expert
* Any ongoing medication impacting the postprandial glucose and insulin response (like beta blockers), to the opinion of the medical expert
* Any ongoing medication impacting brain metabolism or function (neuroleptics, antidepressants, anti-epileptics), to the opinion of the medical expert
* Ongoing chemotherapy
* Any food supplement intake (e.g. MCT, ketone salts = Calcium, Sodium, Potassium, Magnesium) or special diet (e.g. ketogenic diet) possibly impacting basal ketone levels, to the opinion of the medical expert.
* Claustrophobia
* Hearing disorders (the participant placed into the MRS tunnel should be able to hear from the operators, for safety purpose)
* Having any metallic, electronic, magnetic, or mechanical implants, devices, or objects, for safety reason linked to magnetic field exposure (MRS):

  * Aneurysm clip(s)
  * Cardiac pacemaker
  * Implanted cardioverter defibrillator (ICD)
  * Electronic implant or device
  * Magnetically-activated implant or device
  * Neurostimulation system
  * Spinal cord stimulator
  * Cochlear implant or implanted hearing aid
  * Insulin or infusion pump
  * Implanted drug infusion device, like portacath® for instance
  * Any type of prosthesis or implant
  * Artificial or prosthetic limb
  * Any metallic fragment or foreign body
  * Hearing aid
  * Other implant
* Subject injured by a metallic object or foreign body
* Allergy to cow milk or soy proteins
* Currently participating or having participated in an investigational trial during the past month
* Subjects not willing and/or not able to comply with scheduled visits and the requirements of the research protocol.
* Subject having a hierarchical link with the investigator or co-investigators.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
The change in brain NAD+/NADH ratio (RX) after the intake of the nutrition products | 31P metabolites and fluxes will be measured during one hour 2 times, one before product intake (control) and the second one 45 min after product intake"

CONTACTS AND LOCATIONS:
Locations (1):
- École Polytechnique Fédérale de Lausanne (EPFL) / Center for Biomedical Imaging (CIBM), Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No